CLINICAL TRIAL: NCT00720980
Title: Granuloma Annulare Treated With Rifampin, Ofloxacin, and Minocycline Combination Therapy
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Other Study IDs: IRB5074
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Granuloma Annulare
Keywords: granuloma annulare, ROM
MeSH Terms: conditions — Granuloma Annulare

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Granuloma annulare is a benign, usually self-limiting, cutaneous dermatosis, which typically presents as asymptomatic, flesh-colored or red papules, frequently arranged in an annular pattern on the distal extremities. Although localized granuloma annulare is most commonly observed, a generalized or disseminated form can occur. The etiology of granuloma annulare is unknown, however, multiple inciting factors have been proposed. The purpose of the investigators is to review the outcomes of treatment of granuloma annulare (GA) resistant to standard regimens that resolved after a 3-months treatment course of monthly rifampin, ofloxacin, and minocycline (ROM) therapy, successfully used to treat paucibacillary leprosy, a disease with clinical and histopathologic similarity to GA.

DETAILED DESCRIPTION:
We will document the regimen treatment each patient has had and then review the following from the patient's chart to target our specific aims as outlined above.

1. What previous treatment options have been or/are currently being used?
2. How long did the patient take the treatment for?
3. Was the patient able to discontinue or become less dependent on prior treatment?
4. Was the disease process slowed by the treatment?;
5. Were there any side effects that the patient experienced with treatment?

ELIGIBILITY:
Inclusion Criteria:

* Patients with granuloma annulare who are resistent to the standard treatment.

Exclusion Criteria:

* Response to the standard treatment of granuloma annulare.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators reported 6 cases of resistant GA that resolved after a 3-month treatment course of monthly rifampin, ofloxacin, and minocycline (ROM) therapy. ROM therapy has been successfully used to treat patients with paucibacillary leprosy, which has morphologic and histologic similarities to GA.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2008-05; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H Hamzavi, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Medical Center, Detroit, Michigan, United States

REFERENCES:
- [Background] Duarte AF, Mota A, Pereira MA, Baudrier T, Azevedo F. Generalized granuloma annulare--response to doxycycline. J Eur Acad Dermatol Venereol. 2009 Jan;23(1):84-5. doi: 10.1111/j.1468-3083.2008.02707.x. Epub 2008 Apr 1. No abstract available. PMID 18384540